CLINICAL TRIAL: NCT05235243
Title: Can Mindfulness Meditation and Self-monitoring Can Help Improve Control Over Maladaptive Daydreaming: A Randomized Controlled Trial of a Self-guided Web-based Program
Brief Title: Can Mindfulness and Self-monitoring Improve Control Over Maladaptive Daydreaming?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Eli Somer, Professor Eli Somer, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 035/18
Record Dates: First submitted 2022-01-19; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Internet-Based Intervention; Psychological Intervention; Intervention Study
Keywords: maladaptive daydreaming; immersive daydreaming; absorption; dissociation; behavioral addiction; compulsive behavior; RCT
MeSH Terms: conditions — Dissociative Disorders; Compulsive Behavior

STUDY DESIGN:
Intervention Model Description: An RCT in a double-blind setting comparing three groups across three measurement points in time (baseline, post-intervention, and 6-month follow-up)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Full Intervention (FI) group (Experimental): The full intervention (FI) group received a psycho-education module about MD and its addictive behavior mechanism, a motivation enhancement module based on motivational interviewing, mindfulness modules, and self-monitoring modules.
  Interventions: Other: Online therapeutic intervention for maladaptive daydreaming based on mindfulness and self-monitoring
- The partial intervention (PI) group (Active Comparator): The partial intervention (PI) group received an intervention identical to the FI group (a psycho-education module about MD and its addictive behavior mechanism, a motivation enhancement module based on motivational interviewing, mindfulness modules) with the exclusion of the self-monitoring modules.
  Interventions: Other: Online therapeutic intervention for maladaptive daydreaming based on mindfulness
- Waiting List (WL) group (No Intervention): Waiting List (WL) group did not undergo any intervention during the study period. However, WL participants were told that the program will commence in three months. During their waiting time participants were instructed to reduce their daydreaming activity to the best of their ability. Since all participants were recruited for this study from an online support forum (that is not part of this research design), the investigators labeled WL as the Internet Support as Usual (ISAU) group.

INTERVENTIONS:
Other: Online therapeutic intervention for maladaptive daydreaming based on mindfulness and self-monitoring — An 8-weeks internet-based self-guided intervention program, accompanied by e-mail. The content of the intervention and training modules comprised texts, illustrations, explanatory video and audio lectures, as well as interactive worksheets embedded in each week's lesson. Typically, a lesson started with a textual description of its target and duration. Then, participants received a summary of what had been taught thus far, and finally, a novel technique or skill was introduced. Each lesson required about 60 minutes to complete. Users had open access to web pages of previous lessons. Upon completion of each lesson, participants received a list of home assignments to practice during the following week. Our internet-based program featured a notification and download center containing the program's materials and pertinent messages from the researchers.
  Other Names: Maladaptive daydreaming treatment program (MDTP)
  Arms: The Full Intervention (FI) group
Other: Online therapeutic intervention for maladaptive daydreaming based on mindfulness — An 8-weeks internet-based self-guided intervention program, accompanied by e-mail. The content of the intervention and training modules comprised texts, illustrations, explanatory video and audio lectures, as well as interactive worksheets embedded in each week's lesson. Typically, a lesson started with a textual description of its target and duration. Then, participants received a summary of what had been taught thus far, and finally, a novel technique or skill was introduced. Each lesson required about 60 minutes to complete. Users had open access to web pages of previous lessons. Upon completion of each lesson, participants received a list of home assignments to practice during the following week. Our internet-based program featured a notification and download center containing the program's materials and pertinent messages from the researchers.
  Other Names: Maladaptive daydreaming treatment program lite (MDTP)
  Arms: The partial intervention (PI) group

SUMMARY:
Maladaptive daydreaming (MD) is a compulsive form of daydreaming that causes distress and functional impairment among tens of thousands of self-diagnosed sufferers. This is the first controlled treatment trial for MD. The investigators built an internet-based self-help program for MD and tested the effectiveness of mindfulness and self-monitoring in improving control over MD, comparing three groups across three measurement points in time.

DETAILED DESCRIPTION:
Objective: Maladaptive daydreaming (MD) is a compulsive form of daydreaming that causes distress and functional impairment among tens of thousands of self-diagnosed sufferers. This is the first controlled treatment trial for MD. Method: The investigators built an internet-based self-help program for MD and tested the effectiveness of mindfulness and self-monitoring in improving control over MD, compared to internet-based support as usual (waiting-list group). Participants were randomly assigned to three groups and measured across three points in time (baseline, post-intervention, and 6 months follow-up). The investigators measured the change in daydreaming pathology (MDS-16), daydreaming frequency (DDFS), and daydreaming functioning (DWSAS), alongside changes in psychiatric symptoms (BSI), and intervention outcome (OQ). Changes in mindful attention and awareness skills, compliance with program requirements, and feedback to the program were also measured.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* MD diagnosis
* Not being in any concurrent treatment for MD
* English fluent
* Daily access to the internet, and to a device with internet access
* Give informed consent to the study
* Respondents who reported being on a stable dose of medication for at least three months could take part in the study provided that they did not change their dosages while participating in the study.

Exclusion Criteria:

* Age under 18 years
* No MD diagnosis
* In concurrent psychology therapy for MD
* Not fluent in English
* Not having a daily internet access
* Taking medication for less than three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 697 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in maladaptive daydreaming | Baseline, post, and follow-up (8 month total)
  Change in the 16-item Maladaptive Daydreaming Scale (MDS-16) compared to baseline, measured 2 months and 6 months post-intervention. The MDS-16 is the primary self-report scale that gauges maladaptive daydreaming on a 10-point Likert scale. Scores range from 0 to 100, with the mean score of 40 set as an evidence-based cut-off score for clinical-level MD. Higher scores indicate an elevated level of maladaptive daydreaming, hence, a worse outcome.
Change from baseline in daydreaming frequency | Baseline, post, and follow-up (8 month total)
  Change in the Daydreaming Frequency Scale (DDFS) compared to baseline, measured 2 months and 6 months post-intervention. The DDFS is a 12-item subscale of the Imaginal Processes Inventory, gauging reported daydreaming frequency. Items are marked on a 5-point Likert scale. Scores range from 12 to 60. Higher scores indicate an elevated frequency of daydreaming, hence, a worse outcome.
Change from baseline in work and social adjustment | Baseline, post, and follow-up (8 month total)
  Change in the Daydreaming Work and Social Adjustment Scale (DWSAS) compared to baseline, measured 2 months and 6 months post-intervention. The DWSAS is a 6-item measure assessing adjustment and disfunction in relation to daydreaming. Items are ranked on a 9-point Likert scale ranging from 0 to 8. The DWSAS scores range from 0 to 48. A score of 12 or lower indicates "no pathology and disfunction". Scores between 12 and 24 indicate "pathology and impaired function", while scores of 24 or above suggest "severe pathology and impaired function".

SECONDARY OUTCOMES:
Change from baseline in psychiatric symptoms | Baseline, post, and follow-up (8 month total)
  Change in the Brief Symptom Inventory (BSI) compared to baseline, measured 2 months and 6 months post-intervention. The BSI is a 53-item scale rated on a 5-point Likert scale of general psychopathology. The BSI is divided into nine subscales: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, and four additional items. The BSI total score ranges from 0 to 4. Higher scores suggest elevated psychopathology, hence, a worse outcome.
Change from baseline in intervention outcome | Baseline, post, and follow-up (8 month total)
  Change in the Outcome Questionnaire (OQ) from baseline, measured 2 months and 6 months post-intervention. The OQ is a 45-item scale evaluating the quality of mental health care and its outcome featuring three sub-scales: subjective discomfort, interpersonal relations, and social role performance. The OQ scores range from 0 to 180. Higher scores indicate a worse outcome.

OTHER OUTCOMES:
Change from baseline mindful attention awareness | Baseline, post, and follow-up (8 month total)
  Change in the Mindful Attention Awareness Scale (MAAS) from baseline, measured 2 months and 6 months post-intervention. The MAAS assesses awareness and mindful attention and is a common measure in psychological studies of mindfulness training. It gauges the extent to which participants acquired the target mindfulness skill. This is a 15-item, 6-point Likert scale with scores ranging from 15 to 90. Higher scores suggest a higher level of acquired the target mindfulness skills, hence, a better outcome.
The Feedback Questionnaire | Post-intervention, and follow-up (6 month total)
  The Feedback Questionnaire (FBQ) measures the participants' satisfaction with the program and its contents. The FBQ was administered twice: as an immediate post-intervention assessment and, at a 6-month follow-up. The FBQ contains 21 items: 17 of which were ranked on a 5-point Likert scale, and 4 items were optional open questions. This outcome ranked from 1 to 5. Higher scores present more positive feedback to the treatment program, hence, a better outcome.
The Childhood Trauma Questionnaire | Baseline (1 day)
  The Childhood Trauma Questionnaire (CTQ) is a 28-item scale rated on a 5-point Likert scale. The CTQ has five subscales containing five items each: emotional abuse, physical abuse, sexual abuse, emotional neglect, and physical neglect. Each subscale is rated between 5 to 25. The total CTQ scale scores range from 25 to 125. Higher scores represent more childhood trauma, hence, a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Oren Herscu, PhD, Study Chair — School of Social Work, University of Haifa, Israel; Eli Somer, PhD, Study Director — School of Social Work, University of Haifa, Israel; Nirit Soffer-Dudek, PhD, Principal Investigator — Department of Psychology, Ben-Gurion University of the Negev, Israel
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
Non